CLINICAL TRIAL: NCT00156026
Title: Randomized Trial of Immediate Treatment vs. Colposcopic Follow-up for Biopsy-Proven CIN 1
Brief Title: Immediate Treatment vs Colposcopic Follow-up for Biopsy-Proven CIN 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Mark Levine, Ontario Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2000-CIN1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN 1; cervical intraepithelial neoplasia; cervix; cancer; loop electrosurgical excision procedure; LEEP; expectant management; human papilloma virus; HPV; colposcopy
MeSH Terms: conditions — Uterine Cervical Dysplasia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Immediate Treatment - LEEP - Loop electrosurgical excision procedure
  Interventions: Procedure: loop electrosurgical excision procedure (LEEP)
- 2 (No Intervention): Colposcopic Follow-up

INTERVENTIONS:
Procedure: loop electrosurgical excision procedure (LEEP) — 1. loop electrosurgical excision procedure
  Arms: 1

SUMMARY:
This study looks at immediate treatment of a cervix with CIN 1 versus regular six-month follow-up with colposcopy and treatment if CIN 1 progresses.

DETAILED DESCRIPTION:
In women who present with biopsy-proven CIN 1, to compare the management approach of regular colposcopic follow-up and only treating progressive disease using the LEEP, with an approach of immediate treatment using LEEP. The primary outcome is progression to more advanced disease (i.e., CIN 2, CIN 3 or cancer).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will:

  * have documented CIN 1 by histologic assessment as the highest grade lesion present,
  * have the lesion confined to the cervix and completely visualized,
  * be 16 years or older.

Exclusion Criteria:

* any one of the following will be an excluding characteristic:

  * index Pap smear showing CIN 2, CIN 3 or cancer;
  * index Pap smear shows atypical glandular cells of unknown significance, glandular dysplasia, or malignancy requiring immediate investigation;
  * patients with previously identified CIN 1 by biopsy who are already in a colposcopic surveillance program;
  * unsatisfactory colposcopic exam defined as inability to see the extent of the lesion in the endocervical canal or absence of a lesion on the ectocervix but endocervical curettage shows CIN 1;
  * pregnancy;
  * prior therapy for dysplasia including medical (5FU), surgical (Laser, LEEP) or cryotherapy;
  * prior gynecologic cancer;
  * prior pelvic radiation therapy;
  * inability to attend outpatient follow-up visits because of geographic inaccessibility;
  * other malignancies except non-melanoma skin cancer;
  * immunosuppression due to diseases such as AIDS, organ transplantation, or on immunosuppressive medications such as prednisone, imuran or chemotherapy for diseases like systemic lupus;
  * cognitively impaired or otherwise unable to obtain written informed consent;
  * extension of the CIN 1 lesion to vagina or a separate vaginal lesion showing dysplasia;
  * colposcopically visible condyloma outside of the transformation zone;
  * known allergy to local analgesics;
  * clinically evident vaginitis must be treated and resolved prior to entry on the trial;
  * inability to read and respond in English/French;
  * failure to provide informed consent.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2000-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
progression to more advanced disease | 18 months

SECONDARY OUTCOMES:
persistent CIN 1 after 18 months | 18 months
bleeding. | 18 months
predict disease persistence or progression | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Elit, MD, Study Chair — Juravinski Cancer Centre; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Jim Julian, MMath, Principal Investigator — McMaster University, Dept of Clinical Epidemiology & Biostatistics
Locations (10):
- Brazil (2):
  - Universidade Estadual de Campinas, Campinas
  - Instituto Fernandes Figueira - Oswaldo Cruz Foundation, Rio de Janeiro
- Canada (8):
  - B.C. Cancer Agency, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Brantford General Hospital, Brantford, Ontario
  - Hamilton Health Sciences - Henderson Site, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital du Saint-Sacrement, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan